CLINICAL TRIAL: NCT00982644
Title: NN1250-3579: A 52-week Randomised, Controlled, Open Label, Multicentre, Multinational Treat-to-target Trial Comparing the Efficacy and Safety of SIBA and Insulin Glargine, Both Injected Once Daily in Combination With Oral Anti-diabetic Drugs (OAD), in Subjects With Type 2 Diabetes Mellitus Currently Treated With OAD(s) and Qualifying for More Intensified Treatment / NN1250-3643: An Extension Trial to NN1250-3579 Comparing Safety and Efficacy of NN1250 Plus OAD(s) With Insulin Glargine Plus OAD(s) in Type 2 Diabetes (BEGIN™: Once Long)
Brief Title: Comparison of NN1250 Versus Insulin Glargine in Subjects With Type 2 Diabetes
Acronym: BEGIN™
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN1250-3579; 2008-005776-27 (EudraCT Number); U1111-1111-8692 (Other: WHO); 2009-015754-38 (EudraCT Number); U1111-1114-9426 (Other: WHO); NCT01193309 (obsolete NCT alias)
Record Dates: First submitted 2009-09-22; First posted 2009-09-23 (Estimated); Results first posted 2015-11-13 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2016-12

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin degludec; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IDeg OD (Experimental)
  Interventions: Drug: insulin degludec
- IGlar OD (Active Comparator)
  Interventions: Drug: insulin glargine

INTERVENTIONS:
Drug: insulin degludec — Injected subcutaneously (under the skin) once daily. Dose was individually adjusted.
  Arms: IDeg OD
Drug: insulin glargine — Injected subcutaneously (under the skin) once daily. Dose was individually adjusted.
  Arms: IGlar OD

SUMMARY:
This trial is conducted in Europe and the United States of America (USA). The aim of this trial is to compare NN1250 (insulin degludec (IDeg)) with insulin glargine (IGlar) in subjects with type 2 diabetes never treated with insulin followed by the extension trial investigating the long-term safety and tolerability in terms of comparing NN1250 with insulin glargine in subjects with type 2 diabetes.

All oral anti-diabetic drug (OAD) treatment will be discontinued when trial participant enters the main trial (NN1250-3579) with the exception of metformin and dipeptidyl peptidase-IV (DPP-IV) inhibitor treatment (only in countries where DPP-IV inhibitor treatment is approved for combination treatment together with insulin, otherwise DPP-IV inhibitor treatment is also discontinued). Subjects who consent to participate in the extension trial will continue the treatment (NN1250 or insulin glargine + oral antidiabetic drugs (OADs)) to which they were randomly allocated in the 52 week main trial.

The main period is registered internally at Novo Nordisk as NN1250-3579 while the extension period is registered as NN1250-3643.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus
* Treatment with oral antidiabetic drugs (OADs) for at least three months before trial start at an unchanged dose
* HbA1c: 7.0-10.0%
* Body Mass Index (BMI) no higher than 40.0 kg/m^2
* For the extension trial only: Completion of the 52 week treatment period in trial NN1250-3579 (NCT00982644)

Exclusion Criteria:

* Treatment with exenatide or liraglutide within the last 3 months before trial start
* Cardiovascular disease within the last 6 months
* Uncontrolled treated/untreated severe hypertension
* Pregnancy, breast-feeding, the intention of becoming pregnant or not using adequate contraceptive measures
* Cancer and medical history of cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1030 (Actual)
Dates: Start 2009-09; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (173):
- United States (83):
  - Novo Nordisk Investigational Site, Bay Minette, Alabama
  - Novo Nordisk Investigational Site, Birmingham, Alabama
  - Novo Nordisk Investigational Site, Huntsville, Alabama
  - Novo Nordisk Investigational Site, Goodyear, Arizona
  - Novo Nordisk Investigational Site, Anaheim, California
  - Novo Nordisk Investigational Site, Concord, California
  - Novo Nordisk Investigational Site, La Jolla, California
  - Novo Nordisk Investigational Site, Lancaster, California
  - Novo Nordisk Investigational Site, Long Beach, California
  - Novo Nordisk Investigational Site, Los Angeles, California
  - Novo Nordisk Investigational Site, Mission Hills, California
  - Novo Nordisk Investigational Site, National City, California
  - Novo Nordisk Investigational Site, North Hollywood, California
  - Novo Nordisk Investigational Site, Northridge, California
  - Novo Nordisk Investigational Site, Palm Springs, California
  - Novo Nordisk Investigational Site, San Mateo, California
  - Novo Nordisk Investigational Site, Santa Monica, California
  - Novo Nordisk Investigational Site, Spring Valley, California
  - Novo Nordisk Investigational Site, Tarzana, California
  - Novo Nordisk Investigational Site, Tustin, California
  - Novo Nordisk Investigational Site, Norwalk, Connecticut
  - Novo Nordisk Investigational Site, Boynton Beach, Florida
  - Novo Nordisk Investigational Site, Jacksonville, Florida
  - Novo Nordisk Investigational Site, Melbourne, Florida
  - Novo Nordisk Investigational Site, Miami, Florida
  - Novo Nordisk Investigational Site, New Port Richey, Florida
  - Novo Nordisk Investigational Site, Orange Park, Florida
  - Novo Nordisk Investigational Site, Orlando, Florida
  - Novo Nordisk Investigational Site, Palm Harbor, Florida
  - Novo Nordisk Investigational Site, West Palm Beach, Florida
  - Novo Nordisk Investigational Site, Decatur, Georgia
  - Novo Nordisk Investigational Site, Fort Valley, Georgia
  - Novo Nordisk Investigational Site, Idaho Falls, Idaho
  - Novo Nordisk Investigational Site, Chicago, Illinois
  - Novo Nordisk Investigational Site, Evansville, Indiana
  - Novo Nordisk Investigational Site, Indianapolis, Indiana
  - Novo Nordisk Investigational Site, Lexington, Kentucky
  - Novo Nordisk Investigational Site, Paducah, Kentucky
  - Novo Nordisk Investigational Site, Metairie, Louisiana
  - Novo Nordisk Investigational Site, Slidell, Louisiana
  - Novo Nordisk Investigational Site, Greenbelt, Maryland
  - Novo Nordisk Investigational Site, North East, Maryland
  - Novo Nordisk Investigational Site, Reisterstown, Maryland
  - Novo Nordisk Investigational Site, Rockville, Maryland
  - Novo Nordisk Investigational Site, Brockton, Massachusetts
  - Novo Nordisk Investigational Site, North Dartmouth, Massachusetts
  - Novo Nordisk Investigational Site, St Louis, Missouri
  - Novo Nordisk Investigational Site, Henderson, Nevada
  - Novo Nordisk Investigational Site, Las Vegas, Nevada
  - Novo Nordisk Investigational Site, Toms River, New Jersey
  - Novo Nordisk Investigational Site, Northport, New York
  - Novo Nordisk Investigational Site, Staten Island, New York
  - Novo Nordisk Investigational Site, Asheboro, North Carolina
  - Novo Nordisk Investigational Site, Charlotte, North Carolina
  - Novo Nordisk Investigational Site, Cincinnati, Ohio
  - Novo Nordisk Investigational Site, Dayton, Ohio
  - Novo Nordisk Investigational Site, Toledo, Ohio
  - Novo Nordisk Investigational Site, Oklahoma City, Oklahoma
  - Novo Nordisk Investigational Site, Kingston, Pennsylvania
  - Novo Nordisk Investigational Site, Langhorne, Pennsylvania
  - Novo Nordisk Investigational Site, Melrose Park, Pennsylvania
  - Novo Nordisk Investigational Site, Pittsburgh, Pennsylvania
  - Novo Nordisk Investigational Site, West Reading, Pennsylvania
  - Novo Nordisk Investigational Site, East Providence, Rhode Island
  - Novo Nordisk Investigational Site, Columbia, South Carolina
  - Novo Nordisk Investigational Site, Greer, South Carolina
  - Novo Nordisk Investigational Site, Newberry, South Carolina
  - Novo Nordisk Investigational Site, Chattanooga, Tennessee
  - Novo Nordisk Investigational Site, Harriman, Tennessee
  - Novo Nordisk Investigational Site, Humboldt, Tennessee
  - Novo Nordisk Investigational Site, Nashville, Tennessee
  - Novo Nordisk Investigational Site, Arlington, Texas
  - Novo Nordisk Investigational Site, Corpus Christi, Texas
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, El Paso, Texas
  - Novo Nordisk Investigational Site, Hurst, Texas
  - Novo Nordisk Investigational Site, Irving, Texas
  - Novo Nordisk Investigational Site, Lubbock, Texas
  - Novo Nordisk Investigational Site, San Antonio, Texas
  - Novo Nordisk Investigational Site, Sugar Land, Texas
  - Novo Nordisk Investigational Site, Richmond, Virginia
  - Novo Nordisk Investigational Site, Spokane, Washington
  - Novo Nordisk Investigational Site, Milwaukee, Wisconsin
- Austria (4):
  - Novo Nordisk Investigational Site, Bregenz
  - Novo Nordisk Investigational Site, Feldkirch
  - Novo Nordisk Investigational Site, Vienna
  - Novo Nordisk Investigational Site, Wolfsberg
- Belgium (4):
  - Novo Nordisk Investigational Site, Brussels
  - Novo Nordisk Investigational Site, Ghent
  - Novo Nordisk Investigational Site, Leuven
  - Novo Nordisk Investigational Site, Liège
- Canada (14):
  - Novo Nordisk Investigational Site, Edmonton, Alberta
  - Novo Nordisk Investigational Site, Coquitlam, British Columbia
  - Novo Nordisk Investigational Site, Winnipeg, Manitoba
  - Novo Nordisk Investigational Site, Mount Pearl, Newfoundland and Labrador
  - Novo Nordisk Investigational Site, St. John's, Newfoundland and Labrador
  - Novo Nordisk Investigational Site, Halifax, Nova Scotia
  - Novo Nordisk Investigational Site, London, Ontario
  - Novo Nordisk Investigational Site, Mississauga, Ontario
  - Novo Nordisk Investigational Site, Ottawa, Ontario
  - Novo Nordisk Investigational Site, Scarborough Village, Ontario
  - Novo Nordisk Investigational Site, Toronto, Ontario
  - Novo Nordisk Investigational Site, Québec, Quebec
  - Novo Nordisk Investigational Site, Saint Romuald, Quebec
  - Novo Nordisk Investigational Site, Saint-Marc-des-Carrieres, Quebec
- Czechia (4):
  - Novo Nordisk Investigational Site, Brno
  - Novo Nordisk Investigational Site, Hradec Králové
  - Novo Nordisk Investigational Site, Pilsen
  - Novo Nordisk Investigational Site, Prague
- Denmark (6):
  - Novo Nordisk Investigational Site, Esbjerg
  - Novo Nordisk Investigational Site, Hillerød
  - Novo Nordisk Investigational Site, Holbæk
  - Novo Nordisk Investigational Site, København S
  - Novo Nordisk Investigational Site, Odense
  - Novo Nordisk Investigational Site, Silkeborg
- Finland (6):
  - Novo Nordisk Investigational Site, Helsinki
  - Novo Nordisk Investigational Site, Joensuu
  - Novo Nordisk Investigational Site, Kerava
  - Novo Nordisk Investigational Site, Lohja
  - Novo Nordisk Investigational Site, Oulu
  - Novo Nordisk Investigational Site, Tampere
- France (7):
  - Novo Nordisk Investigational Site, Le Grau-du-Roi
  - Novo Nordisk Investigational Site, Montigny-lès-Metz
  - Novo Nordisk Investigational Site, Nanterre
  - Novo Nordisk Investigational Site, Nantes
  - Novo Nordisk Investigational Site, Nîmes
  - Novo Nordisk Investigational Site, Saint-denis de La Reunion
  - Novo Nordisk Investigational Site, Vénissieux
- Germany (15):
  - Novo Nordisk Investigational Site, Bad Harzburg
  - Novo Nordisk Investigational Site, Berlin
  - Novo Nordisk Investigational Site, Dormagen
  - Novo Nordisk Investigational Site, Dresden
  - Novo Nordisk Investigational Site, Essen
  - Novo Nordisk Investigational Site, Friedrichsthal
  - Novo Nordisk Investigational Site, Hamburg
  - Novo Nordisk Investigational Site, Hohenmölsen
  - Novo Nordisk Investigational Site, Neuwied
  - Novo Nordisk Investigational Site, Pohlheim
  - Novo Nordisk Investigational Site, Rehburg-Loccum
  - Novo Nordisk Investigational Site, Rehlingen-Siersburg
  - Novo Nordisk Investigational Site, Riesa
  - Novo Nordisk Investigational Site, Saint Ingbert
  - Novo Nordisk Investigational Site, Speyer
- Norway (8):
  - Novo Nordisk Investigational Site, Ålesund
  - Novo Nordisk Investigational Site, Bekkestua
  - Novo Nordisk Investigational Site, Elverum
  - Novo Nordisk Investigational Site, Hamar
  - Novo Nordisk Investigational Site, Kongsvinger
  - Novo Nordisk Investigational Site, Oslo
  - Novo Nordisk Investigational Site, Stavanger
  - Novo Nordisk Investigational Site, Trondheim
- Novo Nordisk Investigational Site, Bayamón, Puerto Rico
- Serbia and Montenegro (4):
  - Novo Nordisk Investigational Site, Belgrade
  - Novo Nordisk Investigational Site, Kragujevac
  - Novo Nordisk Investigational Site, Nis
  - Novo Nordisk Investigational Site, Novi Sad
- Serbia (4):
  - Novo Nordisk Investigational Site, Belgrade
  - Novo Nordisk Investigational Site, Kragujevac
  - Novo Nordisk Investigational Site, Niš
  - Novo Nordisk Investigational Site, Novi Sad
- Slovenia (3):
  - Novo Nordisk Investigational Site, Koper
  - Novo Nordisk Investigational Site, Ljubljana
  - Novo Nordisk Investigational Site, Novo Mesto
- Spain (10):
  - Novo Nordisk Investigational Site, Almería
  - Novo Nordisk Investigational Site, Alzira
  - Novo Nordisk Investigational Site, Antequera
  - Novo Nordisk Investigational Site, Ferrol
  - Novo Nordisk Investigational Site, Gijón
  - Novo Nordisk Investigational Site, Inca
  - Novo Nordisk Investigational Site, Palma de Mallorca
  - Novo Nordisk Investigational Site, Puerto del Rosario
  - Novo Nordisk Investigational Site, Seville
  - Novo Nordisk Investigational Site, Valencia

REFERENCES:
- [Result] Ratner RE, Gough SC, Mathieu C, Del Prato S, Bode B, Mersebach H, Endahl L, Zinman B. Hypoglycaemia risk with insulin degludec compared with insulin glargine in type 2 and type 1 diabetes: a pre-planned meta-analysis of phase 3 trials. Diabetes Obes Metab. 2013 Feb;15(2):175-84. doi: 10.1111/dom.12032. Epub 2012 Dec 3. PMID 23130654
- [Result] Sorli C, Warren M, Oyer D, Mersebach H, Johansen T, Gough SC. Elderly patients with diabetes experience a lower rate of nocturnal hypoglycaemia with insulin degludec than with insulin glargine: a meta-analysis of phase IIIa trials. Drugs Aging. 2013 Dec;30(12):1009-18. doi: 10.1007/s40266-013-0128-2. PMID 24170235
- [Result] Einhorn D, Handelsman Y, Bode BW, Endahl LA, Mersebach H, King AB. PATIENTS ACHIEVING GOOD GLYCEMIC CONTROL (HBA1c <7%) EXPERIENCE A LOWER RATE OF HYPOGLYCEMIA WITH INSULIN DEGLUDEC THAN WITH INSULIN GLARGINE: A META-ANALYSIS OF PHASE 3A TRIALS. Endocr Pract. 2015 Aug;21(8):917-26. doi: 10.4158/EP14523.OR. Epub 2015 Jun 29. PMID 26121451
- [Result] Russell-Jones D, Gall MA, Niemeyer M, Diamant M, Del Prato S. Insulin degludec results in lower rates of nocturnal hypoglycaemia and fasting plasma glucose vs. insulin glargine: A meta-analysis of seven clinical trials. Nutr Metab Cardiovasc Dis. 2015 Oct;25(10):898-905. doi: 10.1016/j.numecd.2015.06.005. Epub 2015 Jun 18. PMID 26232910
- [Result] Vora J, Seufert J, Solberg H, Kinduryte O, Johansen T, Hollander P. Insulin degludec does not increase antibody formation versus insulin glargine: an evaluation of phase IIIa trials. Diabetes Obes Metab. 2016 Jul;18(7):716-20. doi: 10.1111/dom.12621. Epub 2016 Feb 8. PMID 26663320
- [Derived] Rodbard HW, Cariou B, Zinman B, Handelsman Y, Philis-Tsimikas A, Skjoth TV, Rana A, Mathieu C; BEGIN Once Long trial investigators. Comparison of insulin degludec with insulin glargine in insulin-naive subjects with Type 2 diabetes: a 2-year randomized, treat-to-target trial. Diabet Med. 2013 Nov;30(11):1298-304. doi: 10.1111/dme.12303. Epub 2013 Sep 30. PMID 23952326
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 166 sites in 12 countries: Austria (6 sites), Belgium (5 sites), Canada (17 sites), Czech Republic (5 sites), Denmark (6 sites), Finland (6 sites), France (7 sites), Germany (16 sites), Norway (8 sites), Serbia (5 sites), Spain (9 sites) and United States (76 sites). Some subjects did not enrol in the extension period.
Pre-assignment Details: All subjects who completed the 52-week main trial (NN51250-3579, NCT00982644) and when found to be eligible for the extension trial, were offered to participate in the 52-week extension trial (NN1250-3643). The total duration of treatment was up to 104 weeks (52 weeks + 52 weeks).
Groups:
- IDeg OD: Insulin degludec (IDeg) was given subcutaneously (s.c) once daily (OD) with the main evening meal in combination with metformin with or without DPP-IV inhibitors. IDeg was given for 52 weeks in the main period and for another 52 weeks in the extension period.
- IGlar OD: Insulin glargine (IGlar) was given subcutaneously (s.c) once daily (OD), according to the local labelling in combination with metformin with or without DPP-IV inhibitors. IGlar was given for 52 weeks in the main period and for another 52 weeks in the extension period.
Period: Main: Week 0 to 52 (NN1250-3579)
Arm/Group | IDeg OD | IGlar OD
Started | 773 | 257
Full Analysis Set | 773 | 257
Exposed | 766 (7 subjects were withdrawn prior to exposure to trial products) | 257
Completed | 607 | 197
Not Completed | 166 | 60
Not completed — Adverse Event | 20 | 5
Not completed — Lack of Efficacy | 7 | 2
Not completed — Protocol Violation | 46 | 18
Not completed — Withdrawal criteria | 9 | 5
Not completed — Unclassified | 84 | 30
Period: Extension: Week 53 to 104 (NN1250-3643)
Arm/Group | IDeg OD | IGlar OD
Started | 551 (Fifty-six subjects did not continue into extension trial) | 174 (Twenty-three subjects did not continue into extension trial)
Completed | 505 | 154
Not Completed | 46 | 20
Not completed — Adverse Event | 12 | 5
Not completed — Lack of Efficacy | 3 | 1
Not completed — Protocol Violation | 2 | 4
Not completed — Withdrawal criteria | 6 | 3
Not completed — Unclassified | 23 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IDeg OD | IGlar OD | Total
Number analyzed (Participants) | 773 | 257 | 1030
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.3 (9.7) | 58.7 (9.9) | 59.1 (9.8)
Gender [Count of Participants; unit: Participants]
  Female | 302 | 90 | 392
  Male | 471 | 167 | 638
Glycosylated haemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin] | 8.2 (0.8) | 8.2 (0.8) | 8.2 (0.8)
Fasting plasma glucose (FPG) [Mean (Standard Deviation); unit: mmol/L] | 9.6 (2.6) | 9.7 (2.6) | 9.7 (2.6)

OUTCOME MEASURES:

1. Primary Outcome: Main Trial (Primary Endpoint): Change in Glycosylated Haemoglobin (HbA1c) After 52 Weeks of Treatment
Description: Change from baseline in HbA1c after 52 weeks of treatment
Time Frame: Week 0, Week 52
Population: The full analysis set (FAS) included all randomised subjects and missing data was imputed using last observation carried forward (LOCF).
Measure: Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin
Arm/Group | IDeg OD | IGlar OD
Number analyzed (Participants) | 773 | 257
percentage of glycosylated haemoglobin | -1.06 (1.01) | -1.19 (0.97)

2. Secondary Outcome: Main Trial (Secondary Endpoint): Rate of Confirmed Hypoglycaemic Episodes
Description: Rate of confirmed hypoglycaemic episodes per 100 patient years of exposure (PYE). Confirmed hypoglycaemic episodes consisted of severe hypoglycaemia as well as minor hypoglycaemic episodes. Severe hypoglycaemic episodes are defined as requiring assistance to administer carbohydrate, glucagon, or other resuscitative actions. Minor hypoglycaemic episodes are defined as able to treat her/himself and plasma glucose below 3.1 mmol/L.
Time Frame: Week 0 to Week 52 + 7 days follow up
Population: The safety analysis set (SAS) included all subjects who received at least one dose of the investigational product or its comparator.
Measure: Number; unit: Episodes/100 years of patient exposure
Arm/Group | IDeg OD | IGlar OD
Number analyzed (Participants) | 766 | 257
Episodes/100 years of patient exposure | 152 | 185

3. Primary Outcome: Extension Trial (Primary Endpoint): Rate of Confirmed Hypoglycaemic Episodes
Description: as for outcome 2
Time Frame: Week 0 to Week 104 + 7 days follow up
Population: The SAS included all subjects who received at least one dose of the investigational product or its comparator in the main trial including subjects carried through to the extension trial.
Measure: Number; unit: Episodes/100 years of patient exposure
Arm/Group | IDeg OD | IGlar OD
Number analyzed (Participants) | 766 | 257
Episodes/100 years of patient exposure | 172 | 205

4. Primary Outcome: Extension Trial (Primary Endpoint): Rate of Nocturnal Confirmed Hypoglycaemic Episodes
Description: Rate of confirmed hypoglycaemic episodes per 100 patient years of exposure (PYE). Confirmed hypoglycaemic episodes consisted of severe hypoglycaemia as well as minor hypoglycaemic episodes. Severe hypoglycaemic episodes are defined as requiring assistance to administer carbohydrate, glucagon, or other resuscitative actions. Minor hypoglycaemic episodes are defined as able to treat her/himself and plasma glucose below 3.1 mmol/L. Nocturnal hypoglycaemic episodes are defined as occurring between 00:01 and 05:59 a.m.
Time Frame: Week 0 to Week 104 + 7 days follow up
Population: as for outcome 3
Measure: Number; unit: Episodes/100 years of patient exposure
Arm/Group | IDeg OD | IGlar OD
Number analyzed (Participants) | 766 | 257
Episodes/100 years of patient exposure | 27 | 46

5. Secondary Outcome: Extension Trial (Secondary Endpoint): Change in Glycosylated Haemoglobin (HbA1c) After 104 Weeks of Treatment
Description: Change from baseline in HbA1c after 104 weeks of treatment
Time Frame: Week 0, Week 104
Population: The FAS included all randomised subjects in the main trial including subjects carried through to the extension trial and missing data was imputed using LOCF.
Measure: Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin
Arm/Group | IDeg OD | IGlar OD
Number analyzed (Participants) | 773 | 257
percentage of glycosylated haemoglobin | -0.95 (1.04) | -1.11 (0.99)

6. Secondary Outcome: Main Trial (Secondary Endpoint): Mean of 9-point Self Measured Plasma Glucose Profile (SMPG) at Week 52
Description: Mean of 9-point SMPG at 52 weeks of treatment. Plasma glucose measured: before breakfast, 90 minutes after start of breakfast, before lunch, 90 minutes after start of lunch, before dinner, 90 minutes after start of dinner, bedtime, at 4 am and before breakfast.
Time Frame: Week 52
Population: The FAS included all randomised subjects and missing data was imputed using LOCF. For 126 subjects all 9-point SMPG values were missing.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | IDeg OD | IGlar OD
Number analyzed (Participants) | 681 | 223
mmol/L | 7.7 (1.8) | 7.7 (2.0)

7. Secondary Outcome: Extension Trial (Secondary Endpoint): Mean of 9-point Self Measured Plasma Glucose Profile (SMPG) at Week 104
Description: Mean of 9-point SMPG at 104 weeks of treatment. Plasma glucose measured: before breakfast, 90 minutes after start of breakfast, before lunch, 90 minutes after start of lunch, before dinner, 90 minutes after start of dinner, bedtime, at 4 am and before breakfast.
Time Frame: Week 104
Population: The FAS included all randomised subjects in the main trial including subjects carried through to the extension trial and missing data was imputed using LOCF. For 140 subjects all 9-point SMPG values were missing.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | IDeg OD | IGlar OD
Number analyzed (Participants) | 666 | 224
mmol/L | 7.6 (1.9) | 7.6 (1.9)

8. Secondary Outcome: Main Trial (Secondary Endpoint): Rate of Nocturnal Confirmed Hypoglycaemic Episodes
Description: as for outcome 4
Time Frame: Week 0 to Week 52 + 7 days follow up
Population: The SAS included all subjects who received at least one dose of the investigational product or its comparator.
Measure: Number; unit: Episodes/100 years of patient exposure
Arm/Group | IDeg OD | IGlar OD
Number analyzed (Participants) | 766 | 257
Episodes/100 years of patient exposure | 25 | 39

9. Primary Outcome: Extension Trial (Primary Endpoint): Rate of Treatment Emergent Adverse Events (AEs)
Description: Corresponds to rate of AEs per 100 patient years of exposure. Severity assessed by investigator. Mild: no or transient symptoms, no interference with subject's daily activities. Moderate: marked symptoms, moderate interference with subject's daily activities. Severe: considerable interference with subject's daily activities, unacceptable. Serious AE: AE that at any dose results in any of the following: death, a life-threatening experience, in-subject hospitalization/prolongation of existing hospitalisation, persistent/significant disability/incapacity/congenital anomaly/birth defect.
Time Frame: Week 0 to Week 104 + 7 days of follow up
Population: as for outcome 3
Measure: Number; unit: Events/100 years of patient exposure
Arm/Group | IDeg OD | IGlar OD
Number analyzed (Participants) | 766 | 257
Events/100 years of patient exposure
  Adverse event (AE) | 362 | 339
  Serious AE | 15 | 17
  Severe AE | 14 | 17
  Moderate AE | 93 | 87
  Mild AE | 254 | 234
  Fatal AE | 0 | 1

ADVERSE EVENTS:
Time Frame: Adverse events were collected in a time frame of 104 weeks + 7 days follow up.
Description: The SAS included all subjects who received at least one dose of investigational product or its comparator.
Arm/Group | IDeg OD | IGlar OD
Serious Adverse Events (participants affected / at risk) | 116/766 | 41/257
Other Adverse Events (participants affected / at risk) | 463/766 | 153/257
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDeg OD (N=766) | IGlar OD (N=257)
Acute coronary syndrome (Cardiac disorders) | 4 (4) | 0 (0)
Angina pectoris (Cardiac disorders) | 4 (4) | 2 (3)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 4 (4) | 2 (2)
Atrial flutter (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac failure (Cardiac disorders) | 2 (3) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 3 (4) | 2 (2)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 1 (1)
Congestive cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 10 (11) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 2 (2) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 3 (3) | 2 (2)
Mitral valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 3 (3) | 2 (2)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Tachyarrhythmia (Cardiac disorders) | 2 (2) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (2) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hyperparathyroidism primary (Endocrine disorders) | 1 (1) | 0 (0)
Lens dislocation (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colonic polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 2 (2) | 0 (0)
Hernia (General disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Bronchopneumonia (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Lobar pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 4 (4) | 2 (2)
Pneumonia primary atypical (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Vaginal infection (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Soft tissue injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hypoglycaemic unconsciousness (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder adenocarcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Prostate cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrospinal fistula (Nervous system disorders) | 1 (1) | 0 (0)
Cervicobrachial syndrome (Nervous system disorders) | 2 (2) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 2 (2) | 0 (0)
Syncope (Nervous system disorders) | 3 (3) | 1 (1)
Thalamic infarction (Nervous system disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 2 (2) | 0 (0)
Calculus bladder (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 2 (2) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypertensive crisis (Vascular disorders) | 2 (2) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Acute myocardial ischaemia (Cardiac disorders) | 5 (5) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1
Cardiomyopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Diastolic dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial ishaemia (Cardiac disorders) | 1 (1) | 0 (0)
Sick sinus syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Macular oedema (Eye disorders) | 1 (1) | 0 (0)
Retinal haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enterovesical fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower grastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0) — Cause: Unknown
Multiorgan failure (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis obstructive (Hepatobiliary disorders) | 0 (0) | 1 (1)
Abdominal abscess (Infections and infestations) | 1 (1) | 0 (0)
Diabetic foot (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Meningitis listeria (Infections and infestations) | 0 (0) | 1 (1)
Pseudomembranous colitis (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 0 (0) | 1 (1)
Skin graft infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
In-stent coronary artery restenosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Meniscus lesion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscle injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Diabetic foot (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Rotator cuff syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign neoplasm of prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bronchoalveolar carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon carcinoma stage 3 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Diffuse large B cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Rectal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Renal cell carcinoma stage 1 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebro vascular accident (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (5) | 0 (0)
Embolic cerebral infarction (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hypoglycaemic unconsciousness (Nervous system disorders) | 2 (2) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal cyst (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0)
Urethral stenosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Nasal polyp (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Inguinal hernia repair (Surgical and medical procedures) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDeg OD (N=766) | IGlar OD (N=257)
Diarrhoea (Gastrointestinal disorders) | 83 (126) | 28 (36)
Vomiting (Gastrointestinal disorders) | 34 (44) | 17 (20)
Bronchitis (Infections and infestations) | 70 (99) | 20 (23)
Nasopharyngitis (Infections and infestations) | 183 (310) | 65 (108)
Upper respiratory tract infection (Infections and infestations) | 78 (121) | 19 (33)
Back pain (Musculoskeletal and connective tissue disorders) | 76 (129) | 23 (39)
Headache (Nervous system disorders) | 106 (192) | 30 (57)
Cough (Respiratory, thoracic and mediastinal disorders) | 61 (80) | 14 (20)
Nausea (Gastrointestinal disorders) | 41 (55) | 11 (17)
Oedema peripheral (General disorders) | 46 (55) | 11 (12)
Gastroenteritis (Gastrointestinal disorders) | 34 (40) | 15 (16)
Influenza (Infections and infestations) | 44 (50) | 13 (18)
Urinary tract infection (Infections and infestations) | 45 (64) | 14 (17)
Arthralgia (Musculoskeletal and connective tissue disorders) | 45 (57) | 12 (14)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 30 (37) | 13 (14)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 44 (53) | 11 (11)
Dizziness (Nervous system disorders) | 31 (40) | 14 (18)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk maintains the right to be informed of any Investigator plans for publication and to review any scientific paper, presentation, communication or other information concerning the investigation described in this protocol. Any such communication must be submitted in writing to the Novo Nordisk trial manager prior to submission for comments. Comments will be given within four weeks from receipt of the planned communication.